CLINICAL TRIAL: NCT04137042
Title: Comparison Between 0.9% Saline and Balanced Crystalloid on Intraoperative Metabolomic Profiles Among Patients Undergoing Major Spine Surgery: a Randomized Controlled Trial
Brief Title: Metabolomics of Intraoperative Saline and Balanced Crystalloid Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201907091RINA
Record Dates: First submitted 2019-10-04; First posted 2019-10-23 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2020-11

CONDITIONS: Metabolomics
Keywords: Metabolomics; Fluid therapy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: comparison between two intraoperative iv. fluids
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline (Active Comparator): intraoperative fluid therapy by using 0.9% saline
  Interventions: Drug: Saline
- Balanced crystalloid (Experimental): intraoperative fluid therapy by using balanced crystalloid
  Interventions: Drug: Balanced crystalloid

INTERVENTIONS:
Drug: Saline — Intraoperative fluid therapy is administrated by using 0.9% saline
  Arms: Saline
Drug: Balanced crystalloid — Intraoperative fluid therapy is administrated by using balanced crystalloid
  Arms: Balanced crystalloid

SUMMARY:
Different crystalloids, namely 0.9% saline and balanced crystalloid may result in different metabolomic profile among surgical patients. This study aims to investigate the serum and urine profiles between patients undergoing major spine surgery using 0.9% saline and balanced crystalloid.

DETAILED DESCRIPTION:
Intravenous fluid is mandatory for acute and critically ill patients as well as for surgical patients. Two crystalloid iv. solutions namely 0.9% saline and balanced crystalloid are the most commonly administrated. However, early literature suggests that 0.9% saline is associated with hyperchloremic acidosis, which affects cellular metabolism and may result in worse prognosis among acute or critically ill patients. However, recent literature in 2018, including a meta-analysis and a large randomized controlled trial published in the New England Journal of Medicine revealed neutral or merely slight different clinical outcomes between 0.9% saline and balanced crystalloids. Therefore, the metabolic differences between these two fluids may only exist in specific metabolic pathway which may be easily masked by the complex pathophysiological changes in acute and critically ill patients. These metabolic alteration may be only identified by precise research t the technology such as liquid chromatography mass spectrometry, which provides more comprehensive metabolomics profiles. By comparison, surgical patients undergoing major spine surgery receive a relatively large amount of intravenous infusion during surgery, and there is not complicated with complex pathophysiological alteration of cormorbid diseases. Accordingly, this study aim to identify the metabolomic differences between 0.9% saline and balanced crystalloid among patients undergoing major spine surgery by using the liquid chromatography mass spectrometry technique.

ELIGIBILITY:
Inclusion criteria:

1. age between 40 and 65 year-old
2. major lumbar spine surgery (spinal fusion、multiple levels or expected operation time> 2 hr)

Exclusion criteria:

1. Preoperative organ dysfunction, such as impaired liver function, eg. AST or ALT >100; liver cirrhosis > Child B class; Impaired renal function, eGFR< 60 ml/min/1.73 m2; cardiac dysfunction, such as heart failure > NYHA class II, coronary arterial disease, chronic obstructive pulmonary disease
2. Preoperative use of medications which interfere with liver, renal, glucose or electrolyte metabolism, such as insulin, statin or digoxin
3. Pregnancy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Changes of metabolites in serum and urine measured by metabolomic mass spectrometry | 2-6 hours
  Serum and urine samples will be collected twice (before and immediately after surgery) in each patient.

SECONDARY OUTCOMES:
Intraoperative arterial blood gas profile | 2-6 hours
  Comparison of the arterial blood gas analysis between the two study groups
Intraoperative hemodynamic stability | 2-6 hours
  Comparison of intraoperative norepinephrine requirement between the two study groups

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan